CLINICAL TRIAL: NCT06976255
Title: The Effect of Dark Chocolate and Cinnamon Sugars on Pain and Anxiety in University Students With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: The Effect of Dark Chocolate and Cinnamon Sugars on Pain and Anxiety in University Students With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Principal Investigator, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-SBB-0379
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Primary Dysmenorrhea; Pain; Anxiety
Keywords: university students; dark chocolate; cinnamon sugar
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Dark chocolate (Experimental)
  Interventions: Behavioral: Dark chocolate
- Cinnamon sugar (Experimental)
  Interventions: Behavioral: Cinnamon sugar

INTERVENTIONS:
Behavioral: Cinnamon sugar — In the 2nd and 3rd month of the study, the participants were asked to eat 1 g of cinnamon candies 3 times a day for a total of 4 days, three days before the menstrual cycle and the first day of menstruation.
  Arms: Cinnamon sugar
Behavioral: Dark chocolate — In the 2nd and 3rd month of the study, they were asked to eat 40 mg of 60% cocoa dark chocolate daily for a total of 4 days, three days before the menstrual cycle and the first day of menstruation.
  Arms: Dark chocolate

SUMMARY:
Aim: In this prospective, randomized controlled study, the aim of this study was to investigate the effects of dark chocolate and cinnamon sugar on pain and anxiety in university students with primary dysmenorrhea. Design: The prospective, randomized controlled study

ELIGIBILITY:
Inclusion Criteria:

* University students who had not given birth,
* Were between the ages of 18 and 25,
* Had regular menstrual cycles (28±7 days),
* Had menstrual pain severity of 5 or more on the Visual Analog Scale (VAS) in the previous month,
* Had primary dysmenorrhea, gave written informed consent,
* Volunteered to participate in the study were included in the study.

Exclusion Criteria:

* The study included patients with hearing loss, pelvic pathology, neurological, endocrine or psychiatric disease, and chronic disease such as diabetes mellitus or heart disease, currently taking medication such as antidepressants or oral contraceptives,
* Menstrual irregularities,
* University students who had mental problems that prevented evaluation and cooperation, obesity, malignant condition, pelvic surgery, pregnancy, analgesic use, chocolate and cinnamon allergy,
* Use of any nutritional supplements, medication or non-drug application (reiki, meditation, reflexology, acupressure, etc.) to reduce pain,
* University students who did not volunteer to participate in the study were excluded.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Primary dysmenorrhea
Enrollment: 35 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | change from before implamentation patent and after 1st, 2nd, and 3rd months of practice.]
  The intensity of menstrual pain will be measured using the VAS, a valid and reliable tool for measuring experimental and clinical pain. The VAS is scored on a horizontal line of 10 cm (0=no pain and 10=worst possible pain)
State-Trait Anxiety Inventory | change from before implamentation patent and after 1st, 2nd, and 3rd months of practice.
  There are 40 items in total under two subheadings as State and Trait Anxiety. The Trait Anxiety Scale determines the individual's predisposition to experience anxiety. In the scale consisting of 20 four-point Likert-type questions, items 1, 6, 7, 10, 13, 16, 19 are reverse items. In this scale, a minimum score of 20 and a maximum score of 80 can be obtained. While a high score indicates a high level of anxiety, a low score indicates a low level of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Bartın, Turkey (Türkiye)